CLINICAL TRIAL: NCT04324294
Title: The Role of Contrast Enhanced Endoscopic Ultrasound for Evaluation of Pancreas Lesions
Brief Title: Contrast Enhanced Endoscopic Ultrasound in Pancreas Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Srinivas Gaddam, Assistant Professor of Medicine, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000259
Record Dates: First submitted 2020-03-12; First posted 2020-03-27 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Pancreatitis; Pancreas Cancer; Pancreas Cyst
MeSH Terms: conditions — Pancreatitis; Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Contrast EUS (Experimental): Undergoing EUS for pancreatic indication (cyst, pancreatitis, mass)
  Interventions: Drug: EUS enhanced with contrast to evaluate pancreas

INTERVENTIONS:
Drug: EUS enhanced with contrast to evaluate pancreas — Patients will receive intravenous contrast during EUS to assess whether it improves the evaluation of pancreas.

SUMMARY:
The purpose of this study is to determine whether quantitative contrast-enhanced endoscopic ultrasound (CE-EUS) improves the evaluation of pancreas tumors and precursor lesions, including cysts, compared to conventional endoscopic ultrasound.

DETAILED DESCRIPTION:
The study is a prospective trial of CE- EUS in which the conventional EUS that is part of standard clinical care is conducted after injection of intravenous contrast agent.

The study population will include those patients already undergoing endoscopic ultrasound for standard pancreatic indications at Cedars-Sinai Medical Center. The primary procedures will include conventional EUS to evaluate a pancreatic lesion as part of standard of care, IV contrast agent during the procedure if deemed necessary by the investigator, collection of time intensity curves for pancreas and lesions from the EUS processor. The study includes one standard of care visit for EUS, and the enrollment period will be 24 months. All enrolled patients will be followed by chart review or phone call for a period of 12 months.

All of the subjects will be undergoing an EUS for standard of care. These patients will also receive an IV contrast agent (Lumason) during the procedure, which is not part of standard of care, and is for research use only. FNA will be performed only on those patients deemed to require FNA based solely on the standard EUS.

If the aims of the study are achieved, it ill confirm that contrast-enhanced EUS can be used to differentiate various pancreatic lesions and, in future, may aid in risk-stratification of precursor lesions for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic ultrasound for pancreatic indications
* Patients must have unexplained pancreatitis, pancreas mass(es), or pancreatic cystic lesions or worrisome clinical, imaging or laboratory findings

Exclusion Criteria:

* Patients <18 years of age, pregnant women, and lactating mothers will be excluded.
* Subjects with unstable cardiopulmonary condition will be excluded (acute myocardial infarction, acute coronary syndromes, worsening or unstable heart failure, or serious ventricular arrhythmias)
* Patients with known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts will be excluded given theoretical (though clinically insignificant) risk of embolization
* Patients with a history of allergy to Lumason will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The results obtained by EUS versus contrast EUS to diagnose pancreas cystic lesions, mass lesion, and origin of pancreatitis. | 12 months
  The endoscopist will perform conventional EUS and classify the lesion, which will be recorded by the research assistant prior to CE-EUS. Contrast will then be administered and the classification of CE-EUS will be recorded in real time. Using pathology and one-year clinical follow-up as the gold standard, the yields of the modality will be calculated. In addition, we will evaluate whether the use of CE-EUS impacted assessment of size and diagnosis.

SECONDARY OUTCOMES:
Quantitative Parameters of Pancreas Lesions | 3 months, 6 months, 12 months
  Quantitative parameters of pancreas mass lesions will be performed by comparing the quantitative parameters post processing of adenocarcinoma, other pancreatic lesions, and chronic pancreatitis. The final diagnosis will be based on pathology and 3 , 6 and 12 month follow up. Variables to compare will include time to peak (SECONDS), rise time (SECONDS), mean transit time (SECONDS), and time from peak to one-half (SECONDS).

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Gaddam, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States